CLINICAL TRIAL: NCT03988660
Title: The Circulating Fibrocyte - a Novel and Accurate Biomarker in Diagnosing Acute Appendicitis in Adults
Status: Completed | Type: Observational
Sponsor: University Hospital of Limerick (Other)
Responsible Party: Principal Investigator, Mohamed Zarog, Principal Investigator, University Hospital of Limerick
Other Study IDs: University of Limerick
Record Dates: First submitted 2019-06-11; First posted 2019-06-17 (Actual); Last update posted 2019-06-17 (Actual); Status verified 2019-06

CONDITIONS: Appendicitis
Keywords: Appendicitis; Fibrocytes; Biomarker
MeSH Terms: conditions — Appendicitis | interventions — Lymphocyte Count

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 14 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Healthy controls: Healthy individuals
  Interventions: Diagnostic Test: Circulating fibrocytes
- Histologically confirmed appendicitis: Patients who have diagnosis of appendicitis on histology
  Interventions: Diagnostic Test: Circulating fibrocytes
- Histologically normal appendix: Patients who have diagnosis of a normal appendix on histology
  Interventions: Diagnostic Test: Circulating fibrocytes
- Alternative diagnosis group: Patients who diagnosed with a condition other than appendicitis
  Interventions: Diagnostic Test: Circulating fibrocytes

INTERVENTIONS:
Diagnostic Test: Circulating fibrocytes — Peripheral blood samples were taken from the patients presented with right iliac fossa pain. Samples were collected in sodium heparin (EDTA). Circulating fibrocyte levels were determined by dual staining peripheral blood samples for CD4 and Col-1 using Fluorescence-Activated Cell Sorting (FACS) and correlated with histopathological diagnosis.
  Other Names: White Cell Counts, C-reactive protein, Neutrophils, Lymphocytes, Neutrophil-lymphocyte ratio, Monocytes, Basophils and Eosinophils

SUMMARY:
Accurate diagnostic biomarkers for acute appendicitis (AA) are lacking. Circulating fibrocytes (CFs) are increased in inflammatory states. It is not known whether they are altered in appendicitis. This study aimed to assess if CF altered in AA, and compared their diagnostic accuracy with white cell count (WCC), C-reactive protein (CRP), neutrophils, lymphocytes, neutrophils-lymphocytes ratio (NLR), monocytes, basophils and eosinophils in diagnosis of AA in patients presenting with right iliac fossa pain (RIFP).

95 consecutive adults were recruited in a cohort based prospective study at University Hospital Limerick, 15 were healthy individuals and 80 were patients with RIFP. Peripheral venous samples were obtained at presentation. Clinical, biochemical and histo-pathological parameters were recorded. CF levels were determined by dual-staining for CD45 and Col-1 using FACS and correlated with histopathological diagnoses. P<0.05 was taken as significant.

The study hypothesis is that in patients with suspected appendicitis, CF levels may improve the diagnostics, reduce unnecessary radiation and negative appendicectomy rates.

DETAILED DESCRIPTION:
Acute appendicitis (AA) is the commonest abdominal emergency. Despite its high prevalence, the diagnosis of appendicitis remains a challenge. The clinical presentation is frequently atypical and symptoms often overlap with many other conditions. Coupled with this, failure to reach a prompt diagnosis can result in adverse outcomes.

Circulating fibrocytes (CFs) were first described in 1994 by Richard Bucala. They are haematopoietic cells derived from the bone marrow. They circulate in the monocyte fraction and can differentiate into myelofibrocytes, fibroblasts and adipocytes (among other cell types). They have a prominent role in inflammatory and healing processes, and in the development of fibrosis.

No studies to date have examined the role of CFs in acute appendicitis. Thus, the aims of this clinical trial were (1) to determine if CFs are altered in acute appendicitis, (2) to assess and compare their diagnostic accuracy with CRP, WCC, neutrophils, lymphocytes, neutrophils-lymphocytes ratio (NLR), monocytes, basophils and eosinophils, and (3) to determine the most reliable predictors in diagnosing AA.

A prospective cohort study was undertaken to (1) determine circulating fibrocytes levels (CF) in patients with histologically confirmed acute appendicitis (AA), and (2) to determine the sensitivity and specificity of circulating CF levels in the diagnosis of AA, in adults (age ≥ 16 years) presenting acutely with right iliac fossa pain, at the University hospital Limerick. The diagnosis of appendicitis was confirmed by histopathological assessment following appendicectomy.

Patients were divided in three cohorts following their final diagnosis on discharge and based on the histopathology results. (1) patients with RIFP who underwent an appendicectomy and had a normal appendix at histological assessment i.e histologically proven normal appendix group (HPNG). (2) patients with RIFP who underwent an appendicectomy and had an inflamed appendix at histological assessment i.e histologically proven appendicitis group (HPAG). (3) patients with RIFP who had an alternate diagnosis on discharge other than appendicitis i.e alternative diagnosis group (ADG). Another cohort was added as (4) healthy controls.

Data collected included date of admission, patient's gender, age, presenting symptoms, duration of symptoms, CF levels, preoperative WCC and its differentials (neutrophil, lymphocyte, neutrophils-lymphocytes ratio (NLR), monocyte, basophil and eosinophil counts), CRP, final clinical diagnosis, operation and post-operative diagnosis based at histological assessment.

Peripheral venous samples were obtained from patients in cohort 1, 2 and 3 (n= 80) and healthy controls (n=15). A single 10 mL sample of heparinized venous blood was collected via peripheral, upper extremity venipuncture. Samples were collected in sodium heparin (EDTA) vacutainer tubes and transferred to the laboratory within 3 hours. Samples were then processed to isolate the buffy coat layer using density gradient centrifugation (Histopaque, Sigma-Aldrich, Wicklow, Ireland). The resulting peripheral blood mononuclear cells were subsequently washed in Phosphate-buffered saline (PBS) and re-suspended in freezing medium (50% foetal bovine serum, 40% RPMI medium and 10% dimethyl sulfoxide) prior to transfer to cryogenic vials in 1-ml aliquots. Finally, samples were cooled in a cryogenic temperature control rate container to -80 °C until processing for flow cytometry. Following white blood cell isolation using density gradient centrifugation, 1×106cells were re-suspended in flow cytometry buffer (RPMI medium supplemented with 10% horse serum, 0.1% sodium azide and 25 mM HEPES). Cells were fixed and permeabilised using BD Cytofix/Cytoperm solution (BD Biosciences, Oxford, England) and blocked prior to intracellular staining of Collagen-I with mouse anti-human Collagen-I antibody (Millipore, Cork, Ireland, Product code MAB3391) which was subsequently stained with Alexa-Fluor 488 goat anti-mouse secondary antibody (Jackson ImmunoResearch Europe, Suffolk, England; Product code 115-545-146). Cells were then stained for cell surface antigen CD45 using PerCP anti-human CD45 (Biolegend, London, England). Cells were then re-suspended in PBS before subsequent analysis on the flow cytometer (BD FACSVerse). All analysis was done on a BD FACSVerse (BD Biosciences) using BD FACSuite v1.0.5 (BD Biosciences). Fibrocyte levels were displayed as a percentage of the total white blood cell population.

Data analyses were performed using IBM SPSS for Mac OSX version 25.0. Data were presented as means and standard deviations, or medians and interquartile ranges, as appropriate. Distribution of variables was assessed by histograms, Q-Q plots, and box plots. Analysis of Variance (One-Way ANOVA) was used to compare between different independent groups. Kruskal-Wallis test was used to compare between the biomarkers and the different groups (HPNG vs. HPAG vs. ADG), and for subgroup analysis pairwise comparisons were performed, a P - value of less than 0.05 was considered statistically significant. Receiver operating characteristic (ROC) curve was used to characterize and compare between the diagnostic accuracy of CFs, WCC, CRP, neutrophils, NLR and monocytes. Multinomial logistic regression analysis was used to assess for independent predictors for AA.

ELIGIBILITY:
Inclusion Criteria:

* Any patient presents with right iliac fossa pain
* Age 16 years old or more

Exclusion Criteria:

* Previous appendicectomy

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Healthy individuals and patients presented to the hospital with suspected appendicitis aged 16 year-old- or more.
Sampling Method: Probability Sample
Enrollment: 95 (Actual)
Dates: Start 2015-06-10 (Actual); Primary Completion 2019-04-14 (Actual); Study Completion 2019-04-14 (Actual)

PRIMARY OUTCOMES:
Incidence of patients who have acute appendicitis | 14 days
  The outcome was assessed by histo-pathology analysis post-operatively
Incidence of normal appendix | 14 days
  The outcome was assessed by histo-pathology analysis post-operatively
Incidence of patients with alternative diagnosis | 3 days
  The outcome was assessed clinically following admission

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Limerick, Limerick, Ireland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Zarog M, O'Leary P, Kiernan M, Bolger J, Tibbitts P, Coffey S, Byrnes G, Peirce C, Dunne C, Coffey C. Circulating fibrocyte percentage and neutrophil-lymphocyte ratio are accurate biomarkers of uncomplicated and complicated appendicitis: a prospective cohort study. Int J Surg. 2023 Mar 1;109(3):343-351. doi: 10.1097/JS9.0000000000000234. PMID 37093074